CLINICAL TRIAL: NCT02505594
Title: Pulmonary Vasoreactivity as a Potential Mechanism of Exercise Impairment in Obstructive Sleep Apnea
Brief Title: Potential Mechanism of Exercise Impairment in OSA
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Assistant Professor, University of California, San Diego
Other Study IDs: UCSD150468
Record Dates: First submitted 2015-07-12; First posted 2015-07-22 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Vasoreactivity; Endothelial function; Exercise
MeSH Terms: conditions — Sleep Apnea, Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OSA Group: Apnea-hypopnea index (AHI) ≥ 15 events/h
- Control Group: Apnea-hypopnea index (AHI) < 5 events/h

SUMMARY:
Obstructive sleep apnea (OSA) is a common disorder with major cardiovascular sequelae. A recent study confirmed that OSA is associated with impaired exercise capacity and increasing OSA severity predicts worsening exercise capacity, which is a marker of potential increased cardiovascular risk. However, potential mechanisms of decreased exercise capacity caused by OSA remain unclear. Several pathophysiologic mechanisms of OSA have been proposed and investigators hypothesize that endothelial dysfunction leading to exercise-induced right ventricular dysfunction and associated pulmonary hypertension is the potential mechanism for impaired exercise capacity in OSA.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disorder with major cardiovascular sequelae, including increased systemic hypertension and strokes. OSA is highly prevalent among patients with cardiovascular disease (CVD), but OSA remains under-diagnosed, thus under-treated. Furthermore, a recent study confirmed that OSA is associated with impaired exercise capacity and increasing OSA severity predicts worsening exercise capacity, which is a marker of potential increased cardiovascular risk. However, potential mechanisms of decreased exercise capacity caused by OSA remain unclear.

Several pathophysiologic mechanisms of OSA have been proposed to explain this observation. Endothelial dysfunction is one mechanism that may result from OSA-related intermittent hypoxemia, heightened sympathetic activation, and increased blood pressure. Endothelial dysfunction is characterized by alteration of normal endothelial physiology consisting of a reduction in the bioavailability of vasodilators such as nitric oxide leading to impaired endothelium-depended vasodilation. Endothelial dysfunction has been consistently associated with an increased incidence of CVD. Recent evidence also suggests a correlation between endothelial function and exercise capacity.

In addition, endothelial dysfunction of pulmonary vasculature play an integral role in the pathogenesis of pulmonary hypertension (PH), which is defined by a mean pulmonary artery pressure exceeding 25 mm Hg. PH is associated with increased mortality and multiple morbidities including impaired exercise capacity. OSA has been formally recognized as a cause of PH by the World Health Organization (WHO) and the estimated prevalence of PH in patients with OSA is 17%. Repetitive nocturnal hypoxemia, increased sympathetic tone, and diminished endothelial dependent vaso-reactivity contribute to pulmonary artery hypoxic vasoconstriction, subsequently leading to pulmonary vasculature remodeling and PH. Recently, PH induced by exercise was described as part of the PH spectrum and may represent early, mild, PH that is still clinically relevant in many patients. To detect early PH in OSA patients may signify the importance of treatment and compliance for newly diagnosed OSA patients.

In summary, our hypothesis is that OSA patients may have endothelial dysfunction that leads to impaired exercise capacity via exercise-induced pulmonary hypertension. If our hypothesis is correct, non-invasive measurements of endothelial function could be used clinically to risk stratify patients or follow response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30
* OSA group: diagnosis of untreated moderate-to-severe OSA (apnea-hypopnea index (AHI) ≥ 15 events/h).
* Control group: no OSA (AHI < 5 events/h).

Exclusion Criteria:

* Currently using Continuous Positive Airway Pressure (CPAP) or oral appliance treatment for OSA
* Uncontrolled cardiac co-morbidity, e.g. ischemic heart disease, heart failure, or valvular heart disease that would prevent exercise
* Uncontrolled pulmonary co-morbidity, e.g. asthma or chronic obstructive pulmonary disease (COPD)
* Comorbidities that may severely impair peripheral circulation, e.g. uncontrolled diabetes mellitus, or systemic scleroderma
* Neurological conditions limiting the ability to perform walking or cycling
* Orthopedic condition limiting the ability to perform walking or cycling
* Current smokers, alcohol (> 3 oz/day) or use of illicit drugs.
* Psychiatric disorder, other than mild and controlled depression; e.g. schizophrenia, bipolar disorder, major depression, panic or anxiety disorders.
* Pregnancy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Investigators will enroll 30 subjects with OSA (OSA group) and 30 subjects without OSA (control group). The detailed inclusion and exclusion criteria for subjects are listed below. Female subjects will be offered a urinary pregnancy test and only those documented to be non-pregnant will be studied.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Endothelial function, as measured by endoPAT, between OSA patients and matched healthy controls | Baseline
  EndoPAT is a non-invasive measurement of endothelial function, using peripheral arterial tonometry. Exercise tolerance is measured by Cardiopulmonary exercise testing (CPET). Effects of OSA on exercise tolerance and endothelial function will be evaluated.

SECONDARY OUTCOMES:
Right ventricular systolic pressure (RVSP) in response to exercise | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls
Pulmonary systolic pressure (PASP) in response to exercise | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls
Right ventricular outflow track (RVOT) peak velocity in response to exercise | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls
Velocity time interval (VTI) in response to exercise | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls
Pulmonary artery acceleration time in response to exercise | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls
Systolic peak tricuspid myocardial annular velocity | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls
Diastolic peak tricuspid myocardial annular velocity | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls
Peak tricuspid myocardial annular velocity during isovolumic contraction | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls
Peak tricuspid myocardial annular velocity during isovolumic relaxation | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls
Right ventricular (RV) wall stress | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls
3-D right ventricular ejection fraction (3D-RVEF) | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls
Systolic peak right ventricular (RV) strain | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls
Early diastolic peak right ventricular (RV) strain | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls
Late diastolic peak right ventricular (RV) strain | Baseline
  Measured by Echocardiogram, between OSA patients and matched healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Atul Malhotra, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States